CLINICAL TRIAL: NCT02059863
Title: SPRING (for the Millennium Development Goals): Sustainable Programme Incorporating Nutrition and Games (for Maximising Development, Growth and Survival)
Brief Title: SPRING Cluster Randomised Controlled Trial
Acronym: SPRING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Liverpool (Other); University College, London (Other); Human Development Research Foundation, Pakistan (Other); Sangath (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPNPBE2610; 093615 (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Growth; Stunting, Nutritional; Child Development; Depression, Postpartum; Death
Keywords: cluster randomised trial; low and middle income countries; community based intervention; complex intervention
MeSH Terms: conditions — Growth Disorders; Depression, Postpartum; Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SPRING intervention clusters (Experimental): SPRING package: Home visits by community based agents carried out from pregnancy to 2 years of age to encourage key behaviours to promote child growth, survival and development together with regular supervision
  PLUS access to routine maternal and child health services
  Interventions: Behavioral: SPRING
- Control clusters (No Intervention): access to routine maternal and child health services

INTERVENTIONS:
Behavioral: SPRING — SPRING package: Home visits by community based agents carried out from pregnancy to 2 years of age to encourage key behaviours to promote child growth, survival and development together with regular supervision
  Other Names: Pakistan: Roshan Kal; India: Kilkaari (to be confirmed)
  Arms: SPRING intervention clusters

SUMMARY:
A large number of children in developing countries lack access to known effective interventions. Almost 9 million die each year before reaching their fifth birthday, and over 200 million children who survive fail to achieve their full growth or developmental potential, trapping them in a cycle of continuing disadvantage. The goal of "SPRING", Sustainable Programme Incorporating Nutrition and Games, is to develop an innovative approach to close this access gap, in two of the worst affected countries India and Pakistan, using community based agents. Extensive formative research will be carried out to help ensure that the content and approach of the "SPRING" intervention is feasible, acceptable and appropriately targeted. Findings will be reviewed at an intervention development workshop with local and international stakeholders and experts, and the agreed intervention piloted with a few community based agents and their supervisors. Cluster randomised controlled trials will be carried out in each setting to evaluate the impact of "SPRING" on child growth, development and survival. The programme will include process and economic evaluations to provide information on the total cost of the intervention and its cost effectiveness, as well as development of a framework with lessons learned for implementing "SPRING" in other settings.

DETAILED DESCRIPTION:
The goal of "SPRING", Sustainable Programme Incorporating Nutrition and Games, is to develop an innovative, feasible, affordable and sustainable community based approach that can achieve delivery at scale of known effective interventions that will maximise child development, growth and survival. The vision is to do this by working in close collaboration with government programmes in India and Pakistan, and modifying the approach, content and supervision of existing community based programmes to develop an innovative intervention package that

* Is designed from the outset to be feasible, affordable and appropriate for delivery at scale.
* Is delivered by low cost community based agents through home visits from pregnancy through the first 2 years of life, which

  * promote evidence based newborn and child survival interventions
  * use a problem solving and counselling approach, rather than the standard didactic approach, using techniques informed by evidence from the cognitive behaviour and interpersonal psychotherapy fields.
  * teach care giving skills, such as early recognition of infant signals and capacity, enhancing mother baby interactions, providing stimulation for cognitive growth and development.
  * support optimal infant and young child feeding practices.
  * encourage participation of other family members, e.g. fathers and grandmothers.
  * is informed by the Care for Development Package developed by the World Health Organization (WHO) and the United Nations International Emergency Children's Fund.
* Includes regular supervision, monitoring and evaluation to support the community based agents and ensure the quality of the intervention activities carried out.
* Includes a range of supporting activities developed to provide an enabling environment for mothers and families to carry out the interventions and skills promoted. These might include, for example, community group meetings, and sensitisation sessions with health staff.

The specific objectives of "SPRING" are

1. To test this intervention package through cluster randomised controlled trials in two settings, one in India and one in Pakistan, both with high rates of undernutrition and well established but somewhat different community based agent programmes.
2. To evaluate the impact of the intervention on Infant mortality, child development and growth Maternal psychosocial distress. Coverage of key promoted interventions.
3. To evaluate and monitor all aspects of the intervention process and implementation
4. To cost the delivery of the intervention, and assess its cost effectiveness.
5. To assess the effectiveness of the intervention in reducing inequities in trial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All liveborn babies whose mothers reside within the trial evaluation zones

Exclusion Criteria:

* major congenital malformation
* maternal death in neonatal period

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12000 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
infant mortality | the first year of life
  the % of newborns who die during the first year of life
stunting | 18-24 months
  % children stunted, with stunting defined as below -2 standard deviations of height for age using the WHO growth standards
child development | 18-24 months of age
  a range of psychometric outcome measures covering several domains including cognition, motor, language, and psychosocial development plus maternal-child interaction and quality of the home environment.
maternal psychosocial distress/depression | 6-12 months postpartum
  assessed using the 9 item Patient Health Questionnaire

SECONDARY OUTCOMES:
% adopting key promoted behaviours | from pregnancy up to age 2
wasting | 18-24 months of age
  % children below -2 standard deviations for weight for height using the WHO growth standards.
underweight | 18-24 months of age
  % children below the -2 standard deviations for weight for age using the WHO growth standards.
age-specific infant mortality | during the first year of life
  % babies who die within the following periods after birth: <1 week, 1-3 weeks, 1st month,1-5 months, 6-11 months

CONTACTS AND LOCATIONS:
Overall Officials: Betty Kirkwood, MSc, FMedSci, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- Sangath: Haryana field site, Porvorim, Goa, India
- Human Development Research Foundation: Rawalpindi field site, Islamabad, Punjab Province, Pakistan

REFERENCES:
- [Background] Zafar S, Sikander S, Haq Z, Hill Z, Lingam R, Skordis-Worrall J, Hafeez A, Kirkwood B, Rahman A. Integrating maternal psychosocial well-being into a child-development intervention: the five-pillars approach. Ann N Y Acad Sci. 2014 Jan;1308:107-117. doi: 10.1111/nyas.12339. PMID 24571213
- [Background] Lingam R, Gupta P, Zafar S, Hill Z, Yousafzai A, Iyengar S, Sikander S, Haq ZU, Mehta S, Skordis-Worrel J, Rahman A, Kirkwood B. Understanding care and feeding practices: building blocks for a sustainable intervention in India and Pakistan. Ann N Y Acad Sci. 2014 Jan;1308:204-217. doi: 10.1111/nyas.12326. Epub 2014 Jan 6. PMID 24392960